CLINICAL TRIAL: NCT02349386
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study of BHR-200 (0.36% Transdermal Estradiol Gel) for the Maintenance of Testosterone Suppression in Men With Advanced Androgen-Sensitive Prostate Cancer
Brief Title: Maintaining Suppression of Testosterone With Transdermal Estradiol Gel
Acronym: MASTERS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit patients
Sponsor: BHR Pharma, LLC (Industry)
Collaborators: H2O Clinical LLC (Industry); Q2 Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHR-200-201
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2018-04

CONDITIONS: Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BHR-200 Low Dose (Experimental): 3 mg estradiol per 1 mL 0.36% BHR-200 (transdermal 17β-estradiol gel) applied daily to the skin for up to 52 weeks.
  Interventions: Drug: BHR-200 (0.36% transdermal 17β-estradiol gel)
- BHR-200 Mid Dose (Experimental): 6 mg estradiol per 2 mL 0.36% BHR-200 (transdermal 17β-estradiol gel) applied daily to the skin for up to 52 weeks.
  Interventions: Drug: BHR-200 (0.36% transdermal 17β-estradiol gel)
- BHR-200 High Dose (Experimental): 9 mg estradiol per 3 mL 0.36% BHR-200 (transdermal 17β-estradiol gel) applied daily to the skin for up to 52 weeks.
  Interventions: Drug: BHR-200 (0.36% transdermal 17β-estradiol gel)
- Placebo (Placebo Comparator): 1, 2 or 3 mL of Placebo gel containing 0 mg estradiol applied daily for up to 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHR-200 (0.36% transdermal 17β-estradiol gel) — An absorptive hydroalcoholic gel preparation containing 17β-estradiol.
  Other Names: BHR-200
  Arms: BHR-200 High Dose; BHR-200 Low Dose; BHR-200 Mid Dose
Drug: Placebo — An absorptive hydroalcoholic gel preparation gel of the same ingredients as BHR-200, but without 17β-estradiol.
  Arms: Placebo

SUMMARY:
The objective of this clinical study is to evaluate the safety and efficacy of three different doses of BHR-200 (0.36% transdermal estradiol gel) compared to placebo for the maintenance of testosterone (T) suppression in men with advanced androgen-sensitive prostate cancer.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, dose finding study in men with advanced androgen-sensitive prostate cancer. Patients who give informed consent will have screening evaluations, and if fulfilling the entry criteria, will be randomized to one of 4 treatment groups: 1mL, 2mL or 3mL of 0.36% BHR-200 (transdermal estradiol gel) or Placebo. Study drug will be initiated on the day they were scheduled to receive next depot GnRH agonist injection. Patients will be offered low-dose radiation to aid in the prevention of gynecomastia. Patients will apply the study drug once per day. The first dose of study gel will be applied under the supervision of the PI/designee. Subsequent doses will be self-administered daily by the patient until he is no longer chemically castrated (testosterone levels increase above 50 ng/dL), a rise over baseline PSA of > 0.5 ng/mL is observed, or he has completed 52 weeks of study drug administration. At the conclusion of study participation, patients will be advised to resume standard of care treatment under the supervision of their healthcare provider. While on treatment, patients will be evaluated at Day 1 and every 2 weeks, for the first 24 weeks and every 4 weeks thereafter with a final post-treatment follow-up visit 2 weeks (+/- 1 week) post last dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. Males, Ages 18 and older
2. Body Mass Index (BMI) between 18 and 35 kg/m2 (inclusive)
3. Not currently hospitalized
4. Clinical indication of adenocarcinoma of the prostate evidenced by a biopsy report on record
5. At present receiving ADT treatment with a GnRH agonist for at least 2 months but not longer than 36 months without interruption - Note: If the patient received GnRH agonist treatment prior to the treatment described under 5, there must be evidence of a period without GnRH agonist treatment for a minimum of 2 months prior to starting the present treatment as is seen, for example with intermittent treatment regimens.
6. Able to initiate Screening procedures 2 weeks prior to the next scheduled injection with a GnRH agonist
7. Willing to discontinue current ADT regimen for the duration of the study
8. T level less than 50 ng/dL at Screening
9. WHO/ECOG performance status of 0 or 1
10. Life expectancy of at least 1 year
11. Adequate renal function demonstrated by having normal blood urea nitrogen (BUN) and Creatinine Screening lab values

Exclusion Criteria:

1. History or presence of allergic or adverse response to estradiol
2. Presence of symptomatic metastatic disease, risk of spinal cord compression or urinary obstruction
3. History within the past 2 years of deep vein thrombosis (DVT), pulmonary embolism (PE2), a known thrombophilic disorder (eg.protein C, protein S, or antithrombin deficiency), or cerebrovascular accident (CVA)
4. History within the past 2 years of myocardial infarction or a coronary vascular procedure (e.g. percutaneous coronary intervention, coronary artery bypass graft)
5. History of congestive heart failure
6. Use of any investigational drug, biologic, or device within 28 days prior to the first dose of study gel
7. Use of any of the following known inducers or inhibitors of cytochrome P450 3A4 (CYP3A4): phenobarbital, carbamazepine, rifampin, erythromycin, clarithromycin, ketoconazole, itraconazole, ritonavir, St. John's Wort preparations (Hypericum perforatum), and grapefruit juice
8. Hematological parameters (Hematocrit or Hemoglobin) outside 20% of the upper or lower limits of normal at Screening
9. Active skin rash, sunburn, or other skin disorder on the upper arm(s) that requires treatment or may affect skin absorption of study gel
10. Resting uncontrolled hypertension (HTN) (160/100 mmHg) at Screening
11. Co-existent malignancy or a history of malignancy during the past 5 years, with the exception of basal and/or squamous cell carcinoma of the skin
12. Any other significant concurrent illness or disease or condition that in the opinion of the Investigator might interfere with the patient's ability to receive the treatment outlined in the protocol or might put him at additional risk

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Gerritsen van der Hoop, MD, PhD, Study Director — BHR Pharma, LLC
Locations (12):
- United States (12):
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - South Florida Medical Research, Aventura, Florida
  - Advanced Urology Institute, Daytona Beach, Florida
  - Adult Pediatric Urology, PC, Council Bluffs, Iowa
  - Adult Pediatric Urology, PC, Omaha, Nebraska
  - Delaware Valley Urology, Voorhees Township, New Jersey
  - AccumetRX Clinical Trials, Albuquerque, New Mexico
  - Associated Medical Professionals of NY (AMP of NY), Syracuse, New York
  - Eastern Urological Associates, Greenville, North Carolina
  - Urologic Consultants of Southeastern Pennsylvania (UCSEPA), Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ockrim JL, Lalani EN, Laniado ME, Carter SS, Abel PD. Transdermal estradiol therapy for advanced prostate cancer--forward to the past? J Urol. 2003 May;169(5):1735-7. doi: 10.1097/01.ju.0000061024.75334.40. PMID 12686820
- [Background] Ockrim JL, Lalani el-N, Kakkar AK, Abel PD. Transdermal estradiol therapy for prostate cancer reduces thrombophilic activation and protects against thromboembolism. J Urol. 2005 Aug;174(2):527-33; discussion 532-3. doi: 10.1097/01.ju.0000165567.99142.1f. PMID 16006886
- [Background] Ockrim JL, Abel PD. Long term androgen deprivation therapy in prostate cancer. BMJ. 2008 Sep 22;337:a1361. doi: 10.1136/bmj.a1361. No abstract available. PMID 18809586
- [Background] Ockrim J, Lalani el-N, Abel P. Therapy Insight: parenteral estrogen treatment for prostate cancer--a new dawn for an old therapy. Nat Clin Pract Oncol. 2006 Oct;3(10):552-63. doi: 10.1038/ncponc0602. PMID 17019433
- [Background] Langley RE, Godsland IF, Kynaston H, Clarke NW, Rosen SD, Morgan RC, Pollock P, Kockelbergh R, Lalani el-N, Dearnaley D, Parmar M, Abel PD. Early hormonal data from a multicentre phase II trial using transdermal oestrogen patches as first-line hormonal therapy in patients with locally advanced or metastatic prostate cancer. BJU Int. 2008 Aug;102(4):442-5. doi: 10.1111/j.1464-410X.2008.07583.x. Epub 2008 Apr 16. PMID 18422771
- [Background] Langley RE, Cafferty FH, Alhasso AA, Rosen SD, Sundaram SK, Freeman SC, Pollock P, Jinks RC, Godsland IF, Kockelbergh R, Clarke NW, Kynaston HG, Parmar MK, Abel PD. Cardiovascular outcomes in patients with locally advanced and metastatic prostate cancer treated with luteinising-hormone-releasing-hormone agonists or transdermal oestrogen: the randomised, phase 2 MRC PATCH trial (PR09). Lancet Oncol. 2013 Apr;14(4):306-16. doi: 10.1016/S1470-2045(13)70025-1. Epub 2013 Mar 4. PMID 23465742
- [Background] Bland LB, Garzotto M, DeLoughery TG, Ryan CW, Schuff KG, Wersinger EM, Lemmon D, Beer TM. Phase II study of transdermal estradiol in androgen-independent prostate carcinoma. Cancer. 2005 Feb 15;103(4):717-23. doi: 10.1002/cncr.20857. PMID 15641029
- [Background] Cox RL, Crawford ED. Estrogens in the treatment of prostate cancer. J Urol. 1995 Dec;154(6):1991-8. PMID 7500443
- [Background] Lycette JL, Bland LB, Garzotto M, Beer TM. Parenteral estrogens for prostate cancer: can a new route of administration overcome old toxicities? Clin Genitourin Cancer. 2006 Dec;5(3):198-205. doi: 10.3816/CGC.2006.n.037. PMID 17239273
- [Background] Sayed Y, Taxel P. The use of estrogen therapy in men. Curr Opin Pharmacol. 2003 Dec;3(6):650-4. doi: 10.1016/j.coph.2003.07.004. PMID 14644018

RESULTS

PARTICIPANT FLOW:
Period: 24-Week Double-Blind Main Study
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Started | 9 | 8 | 9 | 8
Completed | 3 | 2 | 4 | 0
Not Completed | 6 | 6 | 5 | 8
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 6 | 6 | 2 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Patient underwent transurethral resection of prostate (exclusionary procedure) | 0 | 0 | 1 | 0
Period: 28-Week Double-Blind Optional Extension
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Started | 3 | 2 | 4 | 0
Completed | 1 | 2 | 1 | 0
Not Completed | 2 | 0 | 3 | 0
Not completed — Lack of Efficacy | 2 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 9 | 8 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 1 | 6
  >=65 years | 7 | 6 | 8 | 7 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 9 | 8 | 9 | 8 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 1 | 1 | 8
  White | 6 | 5 | 8 | 7 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 9 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of Testosterone Suppression at Week 12
Description: Primary Efficacy Endpoint was the percentage of patients failing to maintain castrate levels of T (T < 50 ng/dL).
  Testosterone suppression, defined as the absence of any T level measurement over 50 ng/dL during Weeks 4 to 12.
Time Frame: Week 12
Population: The Intent-to-treat (ITT) population contains all patients who are randomized into the study. All efficacy parameters were analyzed using the ITT population. In the case of a patient who was randomized but did not take the study drug, the analysis was done for this patient using the randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 7
Participants | 3 | 3 | 5 | 2

2. Secondary Outcome: Maintenance of Testosterone Suppression at Week 24
Description: Pproportion of patients failing to maintaincastrate levels of T (T < 50 ng/dL). Testosterone suppression, defined as the absence of any T level measurement over 50 ng/dL during Weeks 4 to 24.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 5 | 6
Participants | 3 | 2 | 3 | 0

3. Secondary Outcome: Number of Patients Reporting Thromboembolic Adverse Events
Description: Number of patients and severity of thromboembolic adverse events
Time Frame: To Week 52/End of Study: Both 24-Week Main Study and Optional 28-Week Extension Study
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 8
Participants | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: Luteinizing Hormone (LH)
Description: Serum concentrations of luteinizing hormone (LH)
Time Frame: Reported for Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Safety population: contains all patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 8
IU/L
  Baseline LH: number analyzed (Participants) | 9 | 8 | 8 | 8
  Baseline LH | 0.380 (0.5700) | 0.470 (0.5949) | 0.190 (0.0000) | 0.530 (0.9576)
  Week 12 LH: number analyzed (Participants) | 3 | 3 | 6 | 2
  Week 12 LH | 0.227 (0.0635) | 0.527 (0.5831) | 1.597 (2.1889) | 2.050 (2.1920)
  Week 24 LH: number analyzed (Participants) | 3 | 2 | 4 | 0
  Week 24 LH | 0.997 (0.7267) | 0.395 (0.2899) | 0.393 (0.4050) |
  Week 36 LH: number analyzed (Participants) | 2 | 2 | 2 | 0
  Week 36 LH | 0.645 (0.6435) | 0.345 (0.2192) | 3.750 (4.7376) |
  Week 48 LH: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 48 LH | 0.600 (0) | 0.300 (0.1414) | 0.300 (0) |

5. Other Pre Specified Outcome: Sex Hormone Binding Globulin (SHBG)
Description: Serum concentrations of sex hormone binding globulin (SHBG)
Time Frame: Reported for Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Safety population: contains all patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 8
nmol/L
  Baseline SHBG: number analyzed (Participants) | 9 | 8 | 8 | 8
  Baseline SHBG | 49.7 (17.65) | 52.8 (22.48) | 45.8 (15.64) | 48.8 (24.09)
  Week 12 SHBG: number analyzed (Participants) | 3 | 3 | 5 | 2
  Week 12 SHBG | 48.7 (18.01) | 55.7 (3.06) | 55.2 (10.62) | 27.0 (2.83)
  Week 24 SHBG: number analyzed (Participants) | 3 | 2 | 3 | 0
  Week 24 SHBG | 50.3 (15.63) | 52.0 (4.24) | 71.3 (8.62) |
  Week 36 SHBG: number analyzed (Participants) | 2 | 2 | 2 | 0
  Week 36 SHBG | 37.0 (7.07) | 53.5 (3.54) | 47.0 (12.73) |
  Week 48 SHBG: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 48 SHBG | 46.0 (0) | 42.5 (7.78) | 58.0 (0) |

6. Other Pre Specified Outcome: Prostate Specific Antigen (PSA)
Description: Serum concentrations of prostate specific antigen (PSA)
Time Frame: To Week 52/End of Study: Both 24-Week Main Study and Optional 28-Week Extension Study
Population: Safety population: contains all patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: ng/ML
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 8
ng/ML
  Baseline PSA: number analyzed (Participants) | 9 | 8 | 8 | 8
  Baseline PSA | 0.374 (0.4572) | 0.921 (1.1726) | 8.058 (22.2814) | 0.334 (0.5623)
  Week 4 PSA: number analyzed (Participants) | 8 | 8 | 8 | 7
  Week 4 PSA | 0.459 (0.6234) | 1.483 (2.2501) | 5.170 (13.1114) | 0.481 (0.6153)
  Week 8 PSA: number analyzed (Participants) | 6 | 4 | 6 | 4
  Week 8 PSA | 0.545 (0.7978) | 1.145 (1.6158) | 4.995 (12.0050) | 0.870 (0.9449)
  Week 12 PSA: number analyzed (Participants) | 3 | 3 | 6 | 2
  Week 12 PSA | 0.330 (0.3251) | 0.227 (0.2367) | 4.380 (10.4936) | 1.395 (1.8455)
  Week 16 PSA: number analyzed (Participants) | 3 | 3 | 3 | 1
  Week 16 PSA | 0.297 (0.2684) | 0.160 (0.1212) | 6.960 (11.8992) | 0.090 (0)
  Week 20 PSA: number analyzed (Participants) | 3 | 3 | 4 | 0
  Week 20 PSA | 0.330 (0.3251) | 0.127 (0.0635) | 5.345 (10.5033) |
  Week 24 PSA: number analyzed (Participants) | 3 | 2 | 4 | 0
  Week 24 PSA | 0.363 (0.3099) | 0.145 (0.0778) | 4.745 (9.3033) |
  Week 28 PSA: number analyzed (Participants) | 3 | 1 | 3 | 0
  Week 28 PSA | 0.430 (0.3110) | 0.090 (0) | 4.863 (8.2590) |
  Week 32 PSA: number analyzed (Participants) | 3 | 2 | 3 | 0
  Week 32 PSA | 0.463 (0.3272) | 0.145 (0.0778) | 4.563 (7.7394) |
  Week 36 PSA: number analyzed (Participants) | 2 | 2 | 2 | 0
  Week 36 PSA | 0.650 (0.0707) | 0.145 (0.0778) | 7.050 (9.5459) |
  Week 40 PSA: number analyzed (Participants) | 2 | 2 | 1 | 0
  Week 40 PSA | 0.750 (0.2121) | 0.145 (0.0778) | 7.800 (0) |
  Week 44 PSA: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 44 PSA | 0.500 (0) | 0.145 (0.0778) | 12.600 (0) |
  Week 48 PSA: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 48 PSA | 0.700 (0) | 0.145 (0.0778) | 12.800 (0) |
  Week 52 PSA: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 52 PSA | 0.700 (0) | 0.145 (0.0778) | 13.300 (0) |

7. Other Pre Specified Outcome: Follicle-stimulating Hormone (FSH)
Description: Serum concentrations of follicle-stimulating hormone (FSH)
Time Frame: Reported for Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Safety population: contains all patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8
IU/L
  Baseline FSH | 4.478 (1.9911) | 5.225 (1.8093) | 3.963 (2.1354) | 5.700 (2.0901)
  Week 12 FSH: number analyzed (Participants) | 3 | 3 | 6 | 2
  Week 12 FSH | 0.630 (0.2339) | 0.493 (0.0058) | 3.848 (5.0343) | 9.450 (5.4447)
  Week 24 FSH: number analyzed (Participants) | 3 | 2 | 4 | 0
  Week 24 FSH | 1.600 (0.9165) | 0.795 (0.4313) | 0.848 (0.5219) |
  Week 36 FSH: number analyzed (Participants) | 2 | 2 | 2 | 0
  Week 36 FSH | 2.050 (1.3435) | 1.095 (0.8556) | 10.600 (12.7279) |
  Week 48 FSH: number analyzed (Participants) | 1 | 2 | 1 | 0
  Week 48 FSH | 2.00 (0) | 0.795 (0.4313) | 1.500 (0) |

8. Other Pre Specified Outcome: Maintenance of Testosterone Suppression at Week 52/ End of Study
Description: Proportion of patients failing to maintain castrate levels of T (T < 50 ng/dL). Testosterone suppression, defined as the absence of any T level measurement over 50 ng/dL during Weeks 24 to 52/End of Study
Time Frame: Double-blind 28-Week Optional Extension Study from Week 24 to Week 52/End of Study
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
Number analyzed (Participants) | 3 | 2 | 4 | 0
Participants | 1 | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: AEs were captured for the duration of the study. The reporting period began with the first dose of Study Drug (Study Day 1) and ends at Week 24 or the End of Study. For participants who opted to enroll in the 28-week open-label extension study, AE collection continued to Week 52 or the End of Study.
Arm/Group | BHR-200 Low Dose | BHR-200 Mid Dose | BHR-200 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 2/9 | 0/8
Other Adverse Events (participants affected / at risk) | 7/9 | 5/8 | 9/9 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BHR-200 Low Dose (N=9) | BHR-200 Mid Dose (N=8) | BHR-200 High Dose (N=9) | Placebo (N=8)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoid tissue operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BHR-200 Low Dose (N=9) | BHR-200 Mid Dose (N=8) | BHR-200 High Dose (N=9) | Placebo (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Application site pain (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 2 | 3 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 1 | 3 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 1 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Nipple disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Lymphoid tissue operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT02349386/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT02349386/SAP_001.pdf